CLINICAL TRIAL: NCT05576662
Title: Selective Trial Of Paxlovid for PASC (STOP-PASC): Randomized Double-Blind Placebo-Controlled Pilot Trial of Paxlovid for the Treatment of PASC
Brief Title: Paxlovid for Treatment of Long Covid
Acronym: STOP-PASC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 66994
Record Dates: First submitted 2022-10-10; First posted 2022-10-12 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Post-acute Sequelae of SARS-CoV-2 Infection; Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — nirmatrelvir; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nirmatrelvir plus ritonavir (Experimental): Participants receive nirmatrelvir plus ritonavir (Paxlovid) for 15 days, and attend follow-up visits through week 15.
  Interventions: Drug: Nirmatrelvir; Drug: Ritonavir
- Placebo plus ritonavir (Placebo Comparator): Participants receive placebo to match nirmatrelvir plus ritonavir for 15 days, and attend follow-up visits through week 15.
  Interventions: Drug: Placebo; Drug: Ritonavir

INTERVENTIONS:
Drug: Nirmatrelvir — Two 150 mg tablets taken by mouth every 12 hours
  Arms: Nirmatrelvir plus ritonavir
Drug: Placebo — Two tablets containing placebo matching nirmatrelvir taken by mouth every 12 hours
  Arms: Placebo plus ritonavir
Drug: Ritonavir — One 100 mg capsule taken by mouth every 12 hours

SUMMARY:
The purpose of this study is to compare whether being treated with nirmatrelvir plus ritonavir for 15 days works better than being treated with placebo plus ritonavir to reduce severe symptoms of Long Covid.

Participants will have 5 planned visits to the study clinic over 15 weeks and will take the drug (or placebo) for the first 15 days.

This study uses the term post-acute sequelae of SARS-CoV-2 (PASC), which is another name for "Long Covid."

DETAILED DESCRIPTION:
An exploratory sub-study will investigate the correlation of physical activity and biometric parameters from digital wearable devices with the subjective symptom severity and other patient-reported outcomes in the main study. All participants with iPhone 6S Plus or newer will be offered an opportunity to opt-in to this sub-study. An Apple Watch and Bluetooth-enabled blood pressure monitor will be provided to participants and data will be collected for the duration of the main study to track participants' physiological and behavioral trends in the Paxlovid versus placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Normal or near-normal kidney function
* History of confirmed COVID-19 infection that preceded the post-COVID symptoms
* Post-COVID-19 symptoms persisting greater than three months
* At least 2 post-COVID symptoms of moderate or severe intensity (fatigue, brain fog, shortness of breath, body aches, gastrointestinal symptoms, or cardiovascular symptoms)
* Willing to report all vaccinations
* Women of childbearing potential or men whose partners may become pregnant must use acceptable method of contraception during the treatment period and for 28 days after the last dose of the study drug
* Willing and able to adhere to study procedures and available for the duration of the study

Exclusion Criteria:

* Suspected or confirmed pregnancy or breastfeeding
* Severe liver disease
* Prior use of study drug or other COVID treatment within 30 days
* Hypersensitivity or other contraindication to any components of the study drug
* Current or expected use of any medication dependent on or inducer of CYP3A4
* Current or expected use of supplements or herbs (unless medically necessary) that cannot be temporarily held (period as determined necessary by investigators)
* HIV infection with viral load >50 copies/ml
* Suspected or confirmed active COVID infection within 30 days
* History of COVID vaccine within 28 days prior to enrollment, or other vaccine (influenza, shingles, etc.) within 14 days of enrollment, or planned use of any vaccine until the primary endpoint has been met (10 weeks)
* Other medical condition(s) or concomitant therapy that would compromise participant's safety or compliance with the study protocol or significantly confound interpretation of study results, as determined by study investigators
* Current enrollment in, or discontinuation within the last 30 days from, a clinical trial involving any investigational drug or device
* Inability to provide informed consent
* Currently hospitalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Upinder Singh, MD, Principal Investigator — Stanford University; Linda Geng, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan for data sharing.

REFERENCES:
- [Result] Geng LN, Bonilla H, Hedlin H, Jacobson KB, Tian L, Jagannathan P, Yang PC, Subramanian AK, Liang JW, Shen S, Deng Y, Shaw BJ, Botzheim B, Desai M, Pathak D, Jazayeri Y, Thai D, O'Donnell A, Mohaptra S, Leang Z, Reynolds GZM, Brooks EF, Bhatt AS, Shafer RW, Miglis MG, Quach T, Tiwari A, Banerjee A, Lopez RN, De Jesus M, Charnas LR, Utz PJ, Singh U. Nirmatrelvir-Ritonavir and Symptoms in Adults With Postacute Sequelae of SARS-CoV-2 Infection: The STOP-PASC Randomized Clinical Trial. JAMA Intern Med. 2024 Sep 1;184(9):1024-1034. doi: 10.1001/jamainternmed.2024.2007. PMID 38848477
- [Result] Gunturkun F, Hedlin H, Botzheim B, Deng Y, Bonilla H, Jagannathan P, Quach TC, Kim S, Lin M, O'Riordan G, Tzeng H, Adamowicz L, Demanuele C, Cai X, Yang PC, Singh U, Geng LN. Digital Biometric Measures in Long COVID: A Secondary Analysis of the STOP-PASC Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2526901. doi: 10.1001/jamanetworkopen.2025.26901. PMID 40810942

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 168 participants were consented and screened. 155 participants were randomized to a study arm.
Groups:
- Nirmatrelvir Plus Ritonavir: Participants receive nirmatrelvir (two 150 mg tablets) plus ritonavir (one 100 mg capsule) every 12 hours for 15 days, and attend follow-up visits through week 15.
- Placebo Plus Ritonavir: Participants receive placebo to match nirmatrelvir plus ritonavir (one 100 mg capsule) every 12 hours for 15 days, and attend follow-up visits through week 15.
Period: Overall Study
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Started | 102 | 53
Completed | 98 | 49
Not Completed | 4 | 4
Not completed — Withdrawn by site within 15-day treatment period | 0 | 1
Not completed — Requested to withdraw within 15-day treatment period | 0 | 1
Not completed — Lost to follow-up within 15-day treatment period | 2 | 0
Not completed — Requested to withdraw after 15-day treatment period | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir | Total
Number analyzed (Participants) | 102 | 53 | 155
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44.5 [35.25 to 56] | 41 [31 to 45] | 43 [34 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 31 | 92
  Male | 41 | 22 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 19
  Not Hispanic or Latino | 90 | 46 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 9 | 20
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 2 | 3
  White | 76 | 39 | 115
  More than one race | 5 | 1 | 6
  Unknown or Not Reported | 8 | 2 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 102 | 53 | 155
Index COVID-19 infection date [Count of Participants; unit: Participants] — Index COVID-19 infection was defined as the initial infection associated with subsequent onset of participant's postacute sequelae of SARS-CoV-2 infection.
  Participants
    Before May 2021 | 39 | 22 | 61
    May to December 2021 | 20 | 7 | 27
    After December 2021 | 43 | 24 | 67
Hospitalized for index COVID-19 infection [Count of Participants; unit: Participants] | 6 | 3 | 9
Time from index infection to randomization [Mean (Standard Deviation); unit: months] | 17.6 (9.1) | 17.3 (9.1) | 17.5 (9.1)
Total COVID-19 infections [Mean (Standard Deviation); unit: infections] — Total COVID-19 infections was the participant-reported total number of COVID-19 infections before enrollment.
  infections | 1.45 (0.75) | 1.34 (0.55) | 1.41 (0.69)
Prior use of SARS-CoV-2 acute medication [Count of Participants; unit: Participants] — Other medications for acute infection include remdesivir, molnupiravir, and bebtelovimab.
  Participants
    Prior use of medication other than Paxlovid | 27 | 14 | 41
    Prior use of Paxlovid | 18 | 9 | 27
    No prior use | 75 | 39 | 114
Vaccination status at randomization [Count of Participants; unit: Participants]
  Initial series completed | 101 | 52 | 153
  Initial series not completed | 1 | 1 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27 (6.19) | 28 (6.66) | 27.55 (6.36)
BMI group [Count of Participants; unit: Participants]
  Underweight (<18.5) | 4 | 0 | 4
  Normal (18.5-24.9) | 39 | 17 | 56
  Overweight (25.0-29.9) | 33 | 18 | 51
  Obesity (≥30.0) | 26 | 18 | 44
Comorbidities [Count of Participants; unit: Participants] — Participant-reported comorbidities included onset before and after the index COVID-19 infection.
  Participants
    Depression | 24 | 13 | 37
    Allergies | 1 | 12 | 13
    Asthma | 15 | 13 | 28
    Anxiety | 15 | 8 | 23
    Gastroesophageal reflux disease (GERD) | 15 | 6 | 21
Moderate to severe post-COVID-19 symptoms [Count of Participants; unit: Participants]
  2-3 symptoms | 47 | 25 | 72
  >3 symptoms | 55 | 28 | 83
Moderate to severe symptom at baseline [Count of Participants; unit: Participants]
  Fatigue | 97 | 51 | 148
  Brain fog | 83 | 42 | 125
  Body aches | 59 | 27 | 86
  Cardiovascular | 50 | 32 | 82
  Shortness of breath | 47 | 28 | 75
  Gastrointestinal | 42 | 25 | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With No, Mild, Moderate, or Severe Symptoms at Week 10 According to the Core Symptoms Severity Scale Score
Description: This measure was to evaluate whether there is a difference between treatment with Paxlovid versus placebo on any of the 6 core symptoms of PASC at week 10 (adjusting for patients' baseline levels). Each symptom (fatigue, brain fog, dyspnea, body aches, gastrointestinal symptoms, cardiovascular symptoms) was assessed on a 4-point Likert scale (range: 0 to 3; 0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms).
Time Frame: Week 10
Population: If participants did not have week 10 data, week 9 data were used when available; otherwise missing data were imputed for statistical analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
Participants
  Fatigue - no symptoms | 3 | 4
  Fatigue - mild symptoms | 22 | 17
  Fatigue - moderate symptoms | 43 | 17
  Fatigue - severe symptoms | 31 | 11
  Brain fog - no symptoms | 11 | 8
  Brain fog - mild symptoms | 34 | 24
  Brain fog - moderate symptoms | 35 | 12
  Brain fog - severe symptoms | 19 | 5
  Dyspnea - no symptoms | 42 | 13
  Dyspnea - mild symptoms | 31 | 21
  Dyspnea - moderate symptoms | 22 | 13
  Dyspnea - severe symptoms | 4 | 2
  Body aches - no symptoms | 31 | 15
  Body aches - mild symptoms | 32 | 17
  Body aches - moderate symptoms | 21 | 14
  Body aches - severe symptoms | 15 | 3
  Gastrointestinal symptoms - no symptoms | 38 | 13
  Gastrointestinal symptoms - mild symptoms | 39 | 17
  Gastrointestinal symptoms - moderate symptoms | 17 | 16
  Gastrointestinal symptoms - severe symptoms | 5 | 3
  Cardiovascular symptoms - no symptoms | 37 | 17
  Cardiovascular symptoms - mild symptoms | 35 | 11
  Cardiovascular symptoms - moderate symptoms | 20 | 13
  Cardiovascular symptoms - severe symptoms | 7 | 8
  Missing Core Symptoms Severity data at week 10 | 3 | 4
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; A proportional odds logistic regression model was fit for severity of each core symptom at week 10, adjusting for baseline severity of the corresponding symptom and fit using only those who experienced the symptom at baseline. A test statistic for overall efficacy was calculated as the weighted average of the treatment coefficient in the proportional odds model for each symptom with inverse variance weighting. The p-value was obtained by a nonparametric permutation test; Test type: Other; p = 0.903, Nonparametric permutation test — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Pooled treatment coefficient = 0.026 — Weighted average of treatment coefficients. A pooled treatment coefficient < 0 favors nirmatrelvir plus ritonavir; a pooled treatment coefficient > 0 favors placebo plus ritonavir

2. Secondary Outcome: Number of Participants With No, Mild, Moderate, or Severe Symptoms at Day 15 According to the Core Symptoms Severity Scale Score
Description: as for outcome 1
Time Frame: Day 15
Population: Participants with symptoms data at day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 99 | 48
Participants
  Fatigue - no symptoms | 3 | 3
  Fatigue - mild symptoms | 17 | 13
  Fatigue - moderate symptoms | 43 | 16
  Fatigue - severe symptoms | 36 | 16
  Brain fog - no symptoms | 7 | 2
  Brain fog - mild symptoms | 36 | 19
  Brain fog - moderate symptoms | 34 | 18
  Brain fog - severe symptoms | 22 | 9
  Dyspnea - no symptoms | 31 | 12
  Dyspnea - mild symptoms | 40 | 20
  Dyspnea - moderate symptoms | 22 | 12
  Dyspnea - severe symptoms | 6 | 4
  Body aches - no symptoms | 21 | 16
  Body aches - mild symptoms | 35 | 15
  Body aches - moderate symptoms | 31 | 13
  Body aches - severe symptoms | 12 | 4
  Gastrointestinal symptoms - no symptoms | 24 | 12
  Gastrointestinal symptoms - mild symptoms | 27 | 14
  Gastrointestinal symptoms - moderate symptoms | 35 | 18
  Gastrointestinal symptoms - severe symptoms | 13 | 4
  Cardiovascular symptoms - no symptoms | 29 | 13
  Cardiovascular symptoms - mild symptoms | 34 | 12
  Cardiovascular symptoms - moderate symptoms | 28 | 13
  Cardiovascular symptoms - severe symptoms | 8 | 10
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of fatigue score at day 15; Test type: Other; p = 0.174, Regression, odds — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Proportional odds regression coefficient Wald test; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.82 to 2.94] — An odds ratio < 1 favors nirmatrelvir plus ritonavir; an odds ratio > 1 favors placebo plus ritonavir
Statistical Analysis 2: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of brain fog score at day 15; Test type: Other; p = 0.548, Regression, odds — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Proportional odds regression coefficient Wald test; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.65 to 2.25] — An odds ratio < 1 favors nirmatrelvir plus ritonavir; an odds ratio > 1 favors placebo plus ritonavir
Statistical Analysis 3: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of dyspnea score at day 15; Test type: Other; p = 0.134, Regression, odds — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Proportional odds regression coefficient Wald test; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.33 to 1.16] — An odds ratio < 1 favors nirmatrelvir plus ritonavir; an odds ratio > 1 favors placebo plus ritonavir
Statistical Analysis 4: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of body aches score at day 15; Test type: Other; p = 0.241, Regression, odds — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Proportional odds regression coefficient Wald test; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.78 to 2.69] — An odds ratio < 1 favors nirmatrelvir plus ritonavir; an odds ratio > 1 favors placebo plus ritonavir
Statistical Analysis 5: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of gastrointestinal symptoms score at day 15; Test type: Other; p = 0.922, Regression, odds — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Proportional odds regression coefficient Wald test; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.55 to 1.92] — An odds ratio < 1 favors nirmatrelvir plus ritonavir; an odds ratio > 1 favors placebo plus ritonavir
Statistical Analysis 6: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of cardiovascular symptoms score at day 15; Test type: Other; p = 0.032, Regression, odds — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Proportional odds regression coefficient Wald test; Odds Ratio (OR) = 0.5, 95% CI 2-sided [0.26 to 0.94] — An odds ratio < 1 favors nirmatrelvir plus ritonavir; an odds ratio > 1 favors placebo plus ritonavir

3. Secondary Outcome: Number of Participants Reporting Relief of at Least One Core Symptom for 2 Weeks
Description: Relief defined as reduction of severity from moderate to none, or severe to mild/none (≥ 2-point Likert score change). Likert score range: 0 to 3; 0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms.
Time Frame: Baseline through week 10, assessed at week 10
Population: Missing data were imputed for statistical analysis, including for participants who were withdrawn prior to week 10
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
Participants | 33 | 22
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Test type: Other; p = 0.09, Regression, Logistic — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Logistic regression coefficient Wald test; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.27 to 1.09] — An odds ratio < 1 favors placebo plus ritonavir; an odds ratio > 1 favors nirmatrelvir plus ritonavir

4. Secondary Outcome: Number of Participants With Overall Alleviation for 2 Weeks
Description: Overall alleviation defined as both:
  1. Any core symptom(s) that are none/mild (Likert 0 or 1) at baseline are none at 10 weeks, and
  2. Any core symptom(s) that are moderate/severe (Likert 2 or 3) at baseline are none/mild at 10 weeks.
  Likert score range: 0 to 3; 0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms.
Time Frame: Baseline through week 10, assessed at week 10
Population: Missing data were imputed for statistical analysis, including for participants who were withdrawn prior to week 10
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
Participants | 7 | 5
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Test type: Other; p = .60, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Logistic regression coefficient Wald test; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.21 to 2.44] — An odds ratio < 1 favors placebo plus ritonavir; an odds ratio > 1 favors nirmatrelvir plus ritonavir

5. Secondary Outcome: Number of Participants With No, Mild, Moderate, or Severe Symptoms of Their Most Bothersome Symptom
Description: This outcome was to assess the severity of the most bothersome symptom experienced by participants. Each symptom was assessed on a 4-point Likert scale (range: 0 to 3; 0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms) using the Core Symptoms Severity Scale.
Time Frame: Assessed at weeks 5, 10, and 15
Population: Missing data were imputed for statistical analysis, including for participants who were withdrawn prior to the respective data collection time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
Participants
  Week 5 - no symptoms | 0 | 1
  Week 5 - mild symptoms | 17 | 12
  Week 5 - moderate symptoms | 41 | 18
  Week 5 - severe symptoms | 34 | 13
  Missing symptoms data at week 5 | 10 | 9
  Week 10 - no symptoms | 3 | 2
  Week 10 - mild symptoms | 22 | 17
  Week 10 - moderate symptoms | 34 | 18
  Week 10 - severe symptoms | 39 | 11
  Missing symptoms data at week 10 | 4 | 5
  Week 15 - no symptoms | 2 | 3
  Week 15 - mild symptoms | 27 | 20
  Week 15 - moderate symptoms | 32 | 17
  Week 15 - severe symptoms | 37 | 7
  Missing symptoms data at week 15 | 4 | 6
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of severity at week 5; Test type: Other; p = 0.156, Regression, odds — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Proportional odds regression coefficient Wald test; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.83 to 3.15] — An odds ratio < 1 favors nirmatrelvir plus ritonavir; an odds ratio > 1 favors placebo plus ritonavir
Statistical Analysis 2: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of severity at week 10; Test type: Other; p = 0.03, Regression, odds — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Proportional odds regression coefficient Wald test; Odds Ratio (OR) = 1.99, 95% CI 2-sided [1.06 to 3.72] — An odds ratio < 1 favors nirmatrelvir plus ritonavir; an odds ratio > 1 favors placebo plus ritonavir
Statistical Analysis 3: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of severity at week 15; Test type: Other; p = 0.01, Regression, odds — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Proportional odds regression coefficient Wald test; Odds Ratio (OR) = 2.42, 95% CI 2-sided [1.27 to 4.60] — An odds ratio < 1 favors nirmatrelvir plus ritonavir; an odds ratio > 1 favors placebo plus ritonavir

6. Secondary Outcome: Time to Relief of the 6 Core Symptoms
Description: Relief defined as reduction of severity from moderate to none, or severe to mild/none for 2 consecutive weeks (≥ 2-point Likert score change). Likert score range: 0 to 3; 0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms.
Time Frame: Up to 15 weeks
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
weeks
  Fatigue | 15 [15 to 15] | 15 [15 to 15]
  Brain fog | 15 [15 to 15] | 15 [15 to 15]
  Body aches | 15 [15 to 15] | 15 [15 to 15]
  Cardiovascular symptoms | 15 [15 to 15] | 15 [15 to 15]
  Shortness of breath | 15 [15 to 15] | 15 [15 to 15]
  Gastrointestinal symptoms | 15 [15 to 15] | 15 [15 to 15]
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of data for "Time to relief - fatigue"; Test type: Other; p = 0.744, Cox PH coefficient Wald test — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.45 to 1.77] — A hazard ratio < 1 favors nirmatrelvir plus ritonavir; a hazard ratio > 1 favors placebo plus ritonavir
Statistical Analysis 2: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of data for "Time to relief - brain fog"; Test type: Other; p = 0.259, Cox PH coefficient Wald test — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.32 to 1.37] — A hazard ratio < 1 favors nirmatrelvir plus ritonavir; a hazard ratio > 1 favors placebo plus ritonavir
Statistical Analysis 3: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of data for "Time to relief - body aches"; Test type: Other; p = 0.286, Cox PH coefficient Wald test — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Hazard Ratio (HR) = 1.61, 95% CI 2-sided [0.65 to 3.99] — A hazard ratio < 1 favors nirmatrelvir plus ritonavir; a hazard ratio > 1 favors placebo plus ritonavir
Statistical Analysis 4: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of data for "Time to relief - cardiovascular symptoms"; Test type: Other; p = 0.846, Cox PH coefficient Wald test — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.38 to 2.24] — A hazard ratio < 1 favors nirmatrelvir plus ritonavir; a hazard ratio > 1 favors placebo plus ritonavir
Statistical Analysis 5: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of data for "Time to relief - shortness of breath"; Test type: Other; p = 0.410, Cox PH coefficient Wald test — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; A hazard ratio < 1 favors nirmatrelvir plus ritonavir; a hazard ratio > 1 favors placebo plus ritonavir; Hazard Ratio (HR) = 1.56, 95% CI 2-sided [0.51 to 4.73]
Statistical Analysis 6: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of data for "Time to relief - gastrointestinal symptoms"; Test type: Other; p = 0.880, Cox PH coefficient Wald test — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.42 to 2.11] — A hazard ratio < 1 favors nirmatrelvir plus ritonavir; a hazard ratio > 1 favors placebo plus ritonavir

7. Secondary Outcome: Time to Relief of the Most Bothersome Symptom
Description: as for outcome 6
Time Frame: Up to 15 weeks
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
weeks | 15 [15 to 15] | 15 [5 to 15]
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Test type: Other; p = 0.33, Cox PH coefficient Wald test — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.40 to 1.38] — A hazard ratio < 1 favors nirmatrelvir plus ritonavir; a hazard ratio > 1 favors placebo plus ritonavir

8. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function T-Score
Description: The PROMIS-Physical Function Short Form (SF) assesses difficulty level performing activities of daily living such as doing chores, climbing stairs, walking, and running errands. The assessment consists of 4 items (questions) with each item scored on 5-point Likert scale (higher scores correspond to better physical function). Scores are computed to a T-score metric, where 50 represents the mean for US general adult population and 10 is the standard deviation. A higher physical function T-score indicates better physical function.
Time Frame: Baseline and week 10
Population: Missing data were imputed for statistical analysis, including for participants who were withdrawn prior to week 10
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
T-score
  Baseline | 37.97 (6.26) | 38.98 (8.71)
  Change at week 10 | 2.73 (6.62) | 1.32 (5.75)
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Test type: Other; p = .66, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Net) = 0.57, 95% CI 2-sided [-1.96 to 3.10] — A mean difference < 0 favors placebo plus ritonavir; a mean difference > 0 favors nirmatrelvir plus ritonavir

9. Secondary Outcome: Change in PROMIS Fatigue T-Score
Description: The PROMIS Fatigue Score assesses level of fatigue and its interference on daily activities. The assessment consists of 7 items (questions) with each item scored on 5-point Likert scale (higher scores correspond to more fatigue). Scores are computed to a T-score metric, where 50 represents the mean for US general adult population and 10 is the standard deviation. A higher fatigue T-score indicates greater fatigue.
Time Frame: Baseline and week 10
Population: Missing data were imputed for statistical analysis, including for participants who were withdrawn prior to week 10
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
T-score
  Baseline | 66.00 (6.42) | 64.00 (6.45)
  Change at week 10 | -3.92 (7.88) | -4.05 (5.90)
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Test type: Other; p = 0.79, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Net) = 0.38, 95% CI 2-sided [-2.40 to 3.15] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir

10. Secondary Outcome: Change in PROMIS Dyspnea-Severity T-Score
Description: The PROMIS-Fatigue Dyspnea-Severity Short Form assesses shortness of breath and its interference on daily activities. The assessment consists of 5 items (questions) scored on 4-point Likert scale with a 7-day recall period (higher scores correspond to worse symptoms). Scores are computed to a T-score metric, where 50 represents the mean for US general adult population and 10 is the standard deviation. A higher Dyspnea-Severity T-score indicates worse symptoms.
Time Frame: Baseline and week 10
Population: Missing data were imputed for statistical analysis, including for participants who were withdrawn prior to week 10
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
T-score
  Baseline | 52.18 (7.49) | 52.59 (8.67)
  Change at week 10 | -1.96 (7.90) | -2.38 (6.13)
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Test type: Other; p = .70, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Net) = 0.60, 95% CI 2-sided [-2.55 to 3.75] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir

11. Secondary Outcome: Change in PROMIS Cognitive Function Abilities T-Score
Description: The PROMIS-Cognitive Function Abilities Short Form assesses brain fog and its interference on daily activities. The assessment consists of 4 items scored on 5-point Likert scale with a 7-day recall period (higher scores indicate better cognitive function). Scores are computed to a T-score metric, where 50 represents the mean for US general adult population and 10 is the standard deviation. A higher Cognitive Function T-score indicates better cognitive function.
Time Frame: Baseline and week 10
Population: Missing data were imputed for statistical analysis, including for participants who were withdrawn prior to week 10
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
T-score
  Baseline | 35.78 (7.90) | 39.09 (6.84)
  Change at week 10 | 4.84 (8.18) | 5.05 (7.56)
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Test type: Other; p = .98, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Net) = 0.03, 95% CI 2-sided [-3.21 to 3.28] — A mean difference < 0 favors placebo plus ritonavir; a mean difference > 0 favors nirmatrelvir plus ritonavir

12. Secondary Outcome: Change in Orthostatic Vitals Test
Description: This outcome measures the difference in supine to standing systolic blood pressure (SBP) and diastolic blood pressure (DBP).
Time Frame: Baseline and week 10
Population: Missing data were imputed for statistical analysis, including for participants who were withdrawn prior to week 10
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Placebo Plus Ritonavir: Participants receive nirmatrelvir (two 150 mg tablets) plus ritonavir (one 100 mg capsule) every 12 hours for 15 days, and attend follow-up visits through week 15.
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
mmHg
  SBP - baseline | 1.79 (12.52) | 3.77 (12.15)
  SBP - change at week 10 | -2.86 (15.9) | -4.47 (14.1)
  DBP - baseline | 6.26 (8.36) | 6.43 (10.90)
  DBP - change at week 10 | -1.86 (1.9) | -1.51 (13.7)
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of data for change of systolic blood pressure; Test type: Other; p = 0.555, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Net) = 1.73, 95% CI 2-sided [-4.06 to 7.53] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir
Statistical Analysis 2: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of data for change of diastolic blood pressure; Test type: Other; p = 0.764, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Net) = -0.68, 95% CI 2-sided [-5.15 to 3.79] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir

13. Secondary Outcome: Change in Heart Rate
Description: This outcome measures the difference in supine to standing heart rate.
Time Frame: Baseline and week 10
Population: Missing data were imputed for statistical analysis, including for participants who were withdrawn prior to week 10
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
bpm
  Baseline | 6.22 (11.92) | 7.70 (8.39)
  Change at week 10 | 0.878 (14.2) | 1.4 (11.5)
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Test type: Other; p = 0.856, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Net) = -0.51, 95% CI 2-sided [-6.15 to 5.12] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir

14. Secondary Outcome: Change in 1-minute Sit-to-stand Test
Description: Number of times participant is able to go from sitting (in an armless chair) to standing in 1 minute (sit to stand cycles).
Time Frame: Baseline and week 10
Population: Missing data were imputed for statistical analysis, including for participants who were withdrawn prior to week 10
Measure: Mean (Standard Deviation); unit: cycles
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
cycles
  Baseline | 20.48 (10.69) | 20.51 (9.80)
  Change at week 10 | 2.67 (10.8) | 3.27 (7.25)
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Test type: Other; p = 0.833, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Net) = -0.41, 95% CI 2-sided [-4.24 to 3.42] — A mean difference < 0 favors placebo plus ritonavir; a mean difference > 0 favors nirmatrelvir plus ritonavir

15. Secondary Outcome: Patient Global Impression of Severity (PGIS) Scale Score
Description: The PGIS reflects a participant's perception about the overall severity of their disease symptoms, rated from 1 to 6 (1 = not present; 2 = very mild; 3 = mild; 4 = moderate; 5 = severe; 6 = extremely severe).
Time Frame: Day 15, and weeks 5, 10, and 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
score on a scale
  Day 15 | 4.04 (0.98) | 3.72 (1.02)
  Week 5 | 4.01 (0.99) | 3.73 (1.02)
  Week 10 | 4.00 (1.03) | 3.79 (1.06)
  Week 15 | 3.94 (1.03) | 3.62 (1.07)
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of day 15 data; Test type: Other; p = 0.096, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.06 to 0.70] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir
Statistical Analysis 2: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of week 5 data; Test type: Other; p = 0.293, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.20 to 0.64] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir
Statistical Analysis 3: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of week 10 data; Test type: Other; p = 0.396, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.25 to 0.62] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir
Statistical Analysis 4: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of week 15 data; Test type: Other; p = 0.064, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-0.02 to 0.77] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir

16. Secondary Outcome: Patient Global Impression of Change (PGIC) Scale Score
Description: The PGIC reflects a participant's perception about the overall efficacy of treatment and their overall status since the start of the treatment, rated from 1 to 7 (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse).
Time Frame: Day 15, and weeks 5, 10, and 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
score on a scale
  Day 15 | 3.74 (1.22) | 3.51 (1.08)
  Week 5 | 3.52 (1.29) | 3.59 (1.13)
  Week 10 | 3.38 (1.31) | 3.13 (1.03)
  Week 15 | 3.38 (1.42) | 3.09 (1.10)
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of day 15 data; Test type: Other; p = 0.444, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.30 to 0.67] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir
Statistical Analysis 2: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of week 5 data; Test type: Other; p = 0.346, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.78 to 0.28] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir
Statistical Analysis 3: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of week 10 data; Test type: Other; p = 0.738, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.48 to 0.67] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir
Statistical Analysis 4: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of week 15 data; Test type: Other; p = 0.578, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.43 to 0.76] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir

17. Secondary Outcome: Summative Severity Score for All Core Symptoms
Description: Core Symptoms Severity Scale Scores for each of the 6 core symptoms were summed to create a summative score. Each core symptom is assessed on a 4-point Likert scale (range: 0 to 3; 0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms). Summative score range: 0 to 18 (high scores correspond to greater severity).
Time Frame: Weeks 5, 10, and 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Nirmatrelvir Plus Ritonavir; Placebo Plus Ritonavir: Participants receive placebo to match nirmatrelvir plus ritonavir (one 100 mg capsule) every 12 hours for 15 days, and attend follow-up visits through week 15.
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
score on a scale
  Week 5: number analyzed (Participants) | 92 | 44
  Week 5 | 8.40 (3.56) | 8.20 (3.88)
  Week 10 | 7.62 (3.75) | 7.69 (4.09)
  Week 15: number analyzed (Participants) | 102 | 47
  Week 15 | 7.90 (3.80) | 7.09 (4.15)
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of week 5 data; Test type: Other; p = 0.758, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-1.41 to 1.03] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir
Statistical Analysis 2: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of week 10 data; Test type: Other; p = 0.693, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-1.46 to 0.97] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir
Statistical Analysis 3: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Analysis of week 15 data; Test type: Other; p = 0.558, Regression, Linear — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Linear regression coefficient Wald test; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-0.87 to 1.61] — A mean difference < 0 favors nirmatrelvir plus ritonavir; a mean difference > 0 favors placebo plus ritonavir

18. Secondary Outcome: Percentage of Weeks 1-15 With Mild or no Symptoms
Description: Each symptom (fatigue, brain fog, dyspnea, body aches, gastrointestinal symptoms, cardiovascular symptoms) is assessed on a 4-point Likert scale (range: 0 to 3; 0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms).
Time Frame: 15 weeks
Population: Missing data were imputed for statistical analysis, including for participants who were withdrawn prior to week 15.
Measure: Median (Inter-Quartile Range); unit: percentage of weeks
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
Number analyzed (Participants) | 102 | 53
percentage of weeks
  Fatigue | 0.15 [0 to 0.39] | 0.15 [0 to 0.77]
  Brain fog | 0.31 [0 to 0.75] | 0.56 [0.15 to 0.85]
  Body Aches | 0.54 [0.10 to 0.92] | 0.64 [0.29 to 0.83]
  Cardiovascular symptoms | 0.67 [0.19 to 0.92] | 0.46 [0 to 0.92]
  Shortness of breath | 0.769 [0.25 to 1] | 0.62 [0.09 to 0.89]
  Gastrointestinal symptoms | 0.63 [0.31 to 0.92] | 0.52 [0.28 to 0.90]
Statistical Analysis 1: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Post-hoc analysis of fatigue data; Test type: Other; p = 0.02, Regression, Logistic — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Logistic regression coefficient Wald test; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.33 to 0.92] — An odds ratio < 1 favors placebo plus ritonavir; an odds ratio > 1 favors nirmatrelvir plus ritonavir
Statistical Analysis 2: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Post-hoc analysis of brain fog data; Test type: Other; p = 0.01, Regression, Logistic — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Logistic regression coefficient Wald test; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.31 to 0.82] — An odds ratio < 1 favors placebo plus ritonavir; an odds ratio > 1 favors nirmatrelvir plus ritonavir
Statistical Analysis 3: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Post-hoc analysis of body aches data; Test type: Other; p = 0.34, Regression, Logistic — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Logistic regression coefficient Wald test; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.74 to 2.33] — An odds ratio < 1 favors placebo plus ritonavir; an odds ratio > 1 favors nirmatrelvir plus ritonavir
Statistical Analysis 4: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Post-hoc analysis of cardiovascular symptoms data; Test type: Other; p = 0.29, Regression, Logistic — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Logistic regression coefficient Wald test; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.76 to 2.48] — An odds ratio < 1 favors placebo plus ritonavir; an odds ratio > 1 favors nirmatrelvir plus ritonavir
Statistical Analysis 5: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Post-hoc analysis of shortness of breath data; Test type: Other; p = 0.35, Regression, Logistic — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Logistic regression coefficient Wald test; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.73 to 2.38] — An odds ratio < 1 favors placebo plus ritonavir; an odds ratio > 1 favors nirmatrelvir plus ritonavir
Statistical Analysis 6: Comparison: Nirmatrelvir Plus Ritonavir vs Placebo Plus Ritonavir; Post-hoc analysis of gastrointestinal symptoms data; Test type: Other; p = 0.25, Regression, Logistic — Uncorrected p-value. A p-value less than the a priori threshold of 0.05 is considered statistically significant; Logistic regression coefficient Wald test; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.79 to 2.47] — An odds ratio < 1 favors placebo plus ritonavir; an odds ratio > 1 favors nirmatrelvir plus ritonavir

ADVERSE EVENTS:
Time Frame: 15 weeks
Arm/Group | Nirmatrelvir Plus Ritonavir | Placebo Plus Ritonavir
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/53
Serious Adverse Events (participants affected / at risk) | 3/102 | 1/53
Other Adverse Events (participants affected / at risk) | 100/102 | 48/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nirmatrelvir Plus Ritonavir (N=102) | Placebo Plus Ritonavir (N=53)
Blood-loss anemia (Blood and lymphatic system disorders) | 1 | 0 — Unrelated to intervention
Forearm fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 — Unrelated to intervention
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Unrelated to intervention
Hepatitis (Hepatobiliary disorders) | 0 | 1 — Possibly related to intervention
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nirmatrelvir Plus Ritonavir (N=102) | Placebo Plus Ritonavir (N=53)
palpitations (Cardiac disorders) | 12 | 7
tachycardia (Cardiac disorders) | 2 | 4
vision blurred (Eye disorders) | 4 | 4
abdominal discomfort (Gastrointestinal disorders) | 9 | 0
abdominal distension (Gastrointestinal disorders) | 6 | 3
abdominal pain (Gastrointestinal disorders) | 21 | 12
constipation (Gastrointestinal disorders) | 9 | 6
diarrhoea (Gastrointestinal disorders) | 51 | 21
dry mouth (Gastrointestinal disorders) | 5 | 3
gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 2
nausea (Gastrointestinal disorders) | 26 | 14
chest pain (General disorders) | 17 | 5
fatigue (General disorders) | 36 | 15
malaise (General disorders) | 6 | 1
pyrexia (General disorders) | 9 | 12
covid-19 (Infections and infestations) | 12 | 5
upper respiratory tract infection (Infections and infestations) | 8 | 2
viral infection (Infections and infestations) | 1 | 6
fibrin d dimer increased (Investigations) | 5 | 3
decreased appetite (Metabolism and nutrition disorders) | 22 | 11
arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 29 | 13
brain fog (Nervous system disorders) | 18 | 9
dizziness (Nervous system disorders) | 17 | 12
dysgeusia (Nervous system disorders) | 63 | 4
headache (Nervous system disorders) | 45 | 13
peripheral sensory neuropathy (Nervous system disorders) | 8 | 5
insomnia (Psychiatric disorders) | 17 | 8
cough (Respiratory, thoracic and mediastinal disorders) | 14 | 7
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 8
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 7
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 13
rash (Skin and subcutaneous tissue disorders) | 6 | 3
hypertension (Vascular disorders) | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT05576662/Prot_SAP_ICF_000.pdf